CLINICAL TRIAL: NCT07030218
Title: A New Red Flag Classification to Predict Vasovagal Syncope During Office Hysteroscopy: A Cross-Sectional Pilot Feasibility Study
Brief Title: A Warning Red Flag Classification System to Predict Risk of Vasovagal Syncope During Office Hysteroscopy
Acronym: FLAG-VS
Status: Enrolling by invitation | Type: Observational
Sponsor: Tanvir Hospital (Other)
Responsible Party: Principal Investigator, Tanvir Singh, Dr, Tanvir Hospital
Other Study IDs: TH/IEC/BHR/0154/2025/TNV/P1/V4
Record Dates: First submitted 2025-05-20; First posted 2025-06-22 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Vasovagal Syncope (VVS)
Keywords: vasovagal syncope; hysteroscopy; red flag classification
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Office hysteroscopy — In office hysteroscopy will utilize 1.9-2.9 mm hysteroscopes (primarily Bettocchi) by the technique of vaginoscopy, without anesthesia or up to level 3a analgesia, in accordance with International Consensus Statement for Recommended Terminology Describing Hysteroscopic Procedures. The choice of distension medium and hysteroscope is left to the operator's discretion. A nurse positioned at the head of the patient will record signs and symptoms of VVR/VVS.

SUMMARY:
The goal of this pilot cross sectional study is to identify participants at risk of vasovagal reaction/syncope(VVR/VVS) during office hysteroscopy. A predictive red flag classification system is being studied to improve procedural safety during office hysteroscopy. Researchers will perform office hysteroscopy as per the standard protocol by vaginoscopic technique. A nurse positioned at the head side of the participant will record signs and symptoms of VVR/VVS. The participant will be asked of the severity of the pain experienced during office hysteroscopy in relation to their menstrual cycle. The procedure will be discontinued at any point the participant wishes to stop.

DETAILED DESCRIPTION:
Office hysteroscopy is increasingly utilized due to advancements in instrumentation and techniques; however, its adoption in routine gynecologic practice remains limited to 10-12% of cases. This under utilization is largely attributed to the perception of pain and lack of financial incentives. Consequently, fewer than 20% of gynecologists employ office hysteroscopy for the evaluation of intrauterine pathology.

Although generally safe, vasovagal syncope (VVS) is the most concerning complication, with a reported prevalence ranging from 0.21% to 1.85%. Other complications include pain, infection, and bleeding. Surgeons often fail to anticipate vasovagal responses during the procedure. This study aims to develop a red flag classification system based on pain response to enable early recognition and prevention of VVS during office hysteroscopy.

Research design This is a multicenter, cross-sectional, analytical pilot study enrolling women undergoing office hysteroscopy over 4 months.

Sample Size Calculation Based on an estimated VVS rate of 6.3%, and using a 95% confidence interval, the sample size of 46 was calculated using Crutzen's online tool.

Statistical Analysis Descriptive analysis will be conducted for continuous and categorical variables. Chi-square tests will evaluate the association between pain classification and vasovagal events. The STROBE checklist will guide reporting.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years
* Prior gynecological care
* Informed consent provided

Exclusion Criteria:

* Inability to consent
* Psychiatric disorders or anxiolytic use
* Use of dilators or anesthesia above level 3a
* Family history of VVS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women undergoing office hysteroscopy in the hospital / outpatient
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of a predictive red flag classification system for identifying patients at risk of vasovagal syncope during office hysteroscopy(OH), with the goal of enhancing procedural safety. | The tolerance level will be assessed perioperative/periprocedural, i.e from the initiation of OH procedure until the completion of the OH procedure.
  During OH, a nurse positioned at the head of the patient will measure and record the tolerance level of the patient at the completion of the procedure using the Red flag Classification:
  Level Description Classification 0 Pain ≤ normal menstruation (Well tolerated) Green Flag
  1. Pain > menstruation, no signs of distress (Tolerated) Green Flag
  2. Level 1 + objective signs (sweating, pallor, malaise) (Tolerated)Red Flag
  3. Level 2 + facial pallor ± loss of consciousness (Not tolerated) Red Flag Normal menstruation is when the pain during periods does not interfere with daily activities. The level of pain tolerated by the women in relation to the menstruation. The feasibility will be assessed by 1) the checking the nurses records which capture the pain scores for any delays or missing data, 2 ) the number of post- procedural pain and tolerance score recorded by the nurse, 3) time taken to complete data 4)Completeness of the data. This information will be used to refine the protocol.

SECONDARY OUTCOMES:
To assess the potential barriers in implementing the red flag classification system, as preparation for a future large-scale validation study | The tolerance level will be assessed perioperative/periprocedural, i.e from the initiation of OH procedure until the completion of the OH procedure.
  The potential barriers are assessed by 1) reviewing the recruitment rate versus the target sample size, 2 ) drop out rate, 3 ) nurses feedback on the ease of recording the tolerance classification, 4) Patient's understanding of the classification and their acceptability to report pain.

OTHER OUTCOMES:
To measure visual analogue score for pain post procedure separately from the tolerance score. | The visual analogue score of pain will be assessed postoperative/postprocedural, i.e immediately after the completion of the OH procedure.
  The visual analogue score for pain is described as - zero which is equivalent to no pain and 10 is the worst possible pain
To measure the body mass index of participant undergoing office hysteroscopy | BMI is calculated when the participant is enrolled in the study to perform office hysteroscopy.
  To measure the weight in kilograms, height in meters, which will be combined to report body mass index (BMI) in kg/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Tanvir Dr., Principal Investigator — Tanvir Hospital
Locations (1):
- Tanvir Hospital, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 2025 -December 2025
Access Criteria: The individual participant data ( IPD ) will be accessible to qualified researchers doing independent scientific research after reviewing the research protocol and statistical analysis plan and execution of data sharing agreement

REFERENCES:
- [Background] Viechtbauer W, Smits L, Kotz D, Bude L, Spigt M, Serroyen J, Crutzen R. A simple formula for the calculation of sample size in pilot studies. J Clin Epidemiol. 2015 Nov;68(11):1375-9. doi: 10.1016/j.jclinepi.2015.04.014. Epub 2015 Jun 6. PMID 26146089
- [Background] Ubeda A, Cabrera S, Escales C, Funes B, Martinez M, Puche A, Martinez Garcia S. Predictors of vasovagal symptoms or syncope during outpatient diagnostic hysteroscopy: A prospective observational study. Eur J Obstet Gynecol Reprod Biol. 2025 May;309:121-125. doi: 10.1016/j.ejogrb.2025.03.044. Epub 2025 Mar 20. PMID 40121697
- [Background] Munro MG, Kasiewicz JL, Desai VB. Office versus Institutional Operative Hysteroscopy: An Economic Model. J Minim Invasive Gynecol. 2022 Apr;29(4):535-548. doi: 10.1016/j.jmig.2021.12.008. Epub 2021 Dec 18. PMID 34933096
- [Background] Isaacson K. Office hysteroscopy: a valuable but under-utilized technique. Curr Opin Obstet Gynecol. 2002 Aug;14(4):381-5. doi: 10.1097/00001703-200208000-00004. PMID 12151827

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT07030218/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-13): https://cdn.clinicaltrials.gov/large-docs/18/NCT07030218/ICF_001.pdf